CLINICAL TRIAL: NCT04761484
Title: A Randomised Trial of Umbilical or Peripheral Catheter Insertion for Preterm Infants on NICU Admission
Brief Title: Umbilical or Peripheral Catheter Insertion for Preterm Infants on Admission to the NICU
Acronym: UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APOLLO_UP
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hypothermia, Newborn; Preterm Birth Complication; Neonatal Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: Randomly assigned in blocks of 4 in a 1:1 ratio, stratified by GA (23 - 25+6, 26 - 28+6) and by admission temperature (normal temperature [36.5oC- 37.5oC] , abnormal temperature [<36.5oC or >37.5oC]).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Insertion of peripheral venous catheter on admission to the NICU
  Interventions: Procedure: Vascular access on admission
- Control (No Intervention): Insertion of and umbilical venous catheter on admission

INTERVENTIONS:
Procedure: Vascular access on admission — PIVC insertion
  Arms: Intervention

SUMMARY:
Preterm infants are at risk of hypothermia following delivery and in the first few hours of life. Hypothermia in extremely low birth weight infants' is an independent risk factor for death. These infants' are at additional risk of hypothermia when they undergo procedures such as central catheter insertion following admission.

The investigators think that in extremely preterm infants, placing a peripheral intravenous cannula on admission to the NICU, instead of umbilical catheters (UVC and/or UAC), will increase the proportion of infants with a rectal temperature in the normal range at 2 hours of life.

DETAILED DESCRIPTION:
Hypothermia is an independent risk factor for death in preterm newborns.(1) Despite measures to improve temperature in preterm newborns in the delivery room (DR), hypothermia on admission to the neonatal intensive care unit (NICU) at NMH is common. In a cohort of infants < 32 weeks' gestation born at NMH in 2019, 54% of infants had a rectal temperature < 36.5 oC on admission to the NICU.(2)

Many preterm infants have procedures performed soon after admission to the NICU; in 2019, 98% of infants born before 29 weeks' gestation at NMH had an umbilical venous catheter inserted. This may/often involve(s) prolonged periods of handling and potential exposure to cold.

The investigators prospectively studied a cohort of 26 infants < 32 weeks who had invasive procedures within 3 hours of birth performed in the NICU at NMH between November 2018 and June 2019. Almost three-quarters [19/26 (73%)] had an abnormal temperature at the beginning of the procedure; and 17/26 (65%) had an abnormal temperature at the end of the procedure. Only 3 (11%) infants maintained a normal temperature throughout the procedure. Perhaps more concerning is the severity of the hypothermia observed; 13 (50%) infants had a temperature < 36.0oC before and 11 (42%) after the procedure. The median duration of procedure was 53 (37, 73) minutes.(3)

The investigators think that in extremely preterm infants, placing a peripheral intravenous cannula on admission to the NICU, instead of umbilical catheters (UVC and/or UAC), will increase the proportion of infants with a rectal temperature in the normal range at 2 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* inborn infants admitted to the NICU with;
* gestational age < 29 weeks (up to 28+6 weeks) OR
* birth weight < 1250g.

Exclusion Criteria:

* end of life (palliative) care
* large abdominal wall defects
* imperforate anus.

Ages: 1 Minute to 60 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Core (rectal) temperature 2 hours after birth | 2 hours
  Core (rectal) temperature 2 hours after birth

SECONDARY OUTCOMES:
Axillary temperature at the end of the procedure | up to 24 hours
Mean difference in axillary temperature from admission to end of procedure | up to 24 hours
Time to completion of procedure (incubator roof down, portholes closed and hands off) | up to 24 hours
Time to first intravenous infusion starting (PN / dextrose / antibiotics / caffeine) | up to 24 hours
Number (%) infants that have umbilical catheters inserted during their admission | up to 24 hours
Number (%) lines used without repositioning | up to 24 hours
Number (%) lines repositioned | up to 24 hours
Number (%) of low lying umbilical venous catheters | up to 24 hours
Number (%) of infants' in whom attempted placement of an umbilical line was not successful | up to 24 hours
  Definition: an attempt made to insert a central catheter that is not used at any point during the infant's admission (i.e. nothing was infused through the line)
Number of peripheral line attempts | up to 24 hours
Number (%) of infants in whom PIVC as first point of access was unsuccessful (nothing was infused through the line) | 24 hours
Complications of line insertion/placement | 10 days
Blood stream infections (CRBSI) | up to 16 weeks
Number of x-rays performed in first 24 hours | 24 hours
Blood sampling in first 24 hours | 24 hours
Number of blood tests in 72 hours | 3 days
Number of blood transfusions during hospital stay | up to 26 weeks
Peripheral arterial line insertion in the first 7 days of life | 7 days
PICC line insertion in the first 7 days of life | 7 days
Inotropes administered in the first 72 hours of life | 3 days
Intubation + Ventilation | Up to 3 days
Surfactant administration | up to 3 days
Necrotizing enterocolitis (Bell's staging) | Up to 3 months
Intraventricular Haemorrhage (Papile classification) | Up to 6 months
Periventricular leukomalacia | Up to 6 months
Chronic lung disease | Up to 3 months
In hospital mortality | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Colm PF O'Donnell, MB BCh BAO, Principal Investigator — The National Maternity Hospital; Lisa K McCarthy, MB BCh BAO, Principal Investigator — The National Maternity Hospital
Locations (1):
- National Maternity Hospital, Dublin, Dubiln, Ireland

IPD SHARING:
Plan to Share IPD: No